CLINICAL TRIAL: NCT06510153
Title: Effect of Live Environmental Music Therapy and Pre-recorded Music on State-Anxiety, Stress, Pain, and Wellbeing Levels of Patients and Caregivers in the Emergency Unit Waiting Area: A Multi-Center Randomized Clinical Trial Study Protocol
Brief Title: Music Therapy and Pre-recorded Music on Patients and Caregivers in the Emergency Unit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Claudia Aristizábal (Other)
Collaborators: Sanitas University (Other)
Responsible Party: Sponsor-Investigator, Claudia Aristizábal, Director, Sanitas University
Organization: Sanitas University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 046-24 UNV
Record Dates: First submitted 2024-07-08; First posted 2024-07-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anxiety; Stress; Well-Being, Psychological
Keywords: Music Therapy; Recorded Music; Anxiety; Stress; Wellbeing; Emergency Care; Waiting Room
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Environmental Music Therapy (Experimental): Environmental Music Therapy (EMT) is a music therapy technique that uses live music to modulate the potentially stressful effects of the environment towards an atmosphere that provides a sense of comfort and security. The instruments used will be an acoustic guitar (Yamaha C-40), an ocean drum (a drum with a double skin on which small metal balls roll imitating the sound of the waves) and a Samafon (an instrument consisting of aluminum tubes of different sizes that are struck with a soft mallet producing long-lasting single or combined tones). The music will consist of improvised music at a slow to moderate tempo, using free-flowing melodies, and simple chord progressions, focusing on creating moments of tension and resolution. The music therapist will also use his/her voice, but without any lyrics or words. After approximately 20 minutes, the music therapist will gradually decrease the volume until the music stops.
  Interventions: Other: Environmental Music Therapy
- Pre-recorded music (Experimental): The protocol for pre-recorded music is the same as for EMT, but instead of using live improvised music, a recording will be used that will consist of the same musical features and musical instruments as the live music. The recording will be made by the same music therapists who will perform the EMT intervention.
  Interventions: Other: Pre-recorded music
- Standard care only (Placebo Comparator): The control group will receive standard care in the emergency room waiting room as provided by each hospital, but without being exposed to EMT or pre-recorded music.
  Interventions: Other: Standard care only

INTERVENTIONS:
Other: Environmental Music Therapy — The music will consist of improvised music at a slow to moderate tempo, using free-flowing melodies, and simple chord progressions, focusing on creating moments of tension and resolution during approximately 20 minutes.
  Arms: Environmental Music Therapy
Other: Pre-recorded music — The protocol for pre-recorded music is the same as for EMT.
  Arms: Pre-recorded music
Other: Standard care only — Standard care in the emergency room waiting room as provided by each hospital without being exposed to EMT or pre-recorded music.
  Arms: Standard care only

SUMMARY:
Patients and caregivers attending emergency units often experience elevated levels of stress and anxiety. Music has been used in waiting rooms to reduce stress and anxiety, but existing studies on music in emergency unit waiting areas are scarce and have limitations such as low statistical power and limited music selection. The aim of this study is to determine the effect of live Environmental Music Therapy (EMT) and pre-recorded music on state-anxiety, stress, pain and well-being levels in patients and caregivers in the emergency unit waiting areas of two hospitals in Colombia.

This study is a multi-center randomized clinical trial, with three arms: standard care + live EMT, standard care + pre-recorded music, and standard care only. The primary outcome measure is the six-item State-Trait Anxiety Inventory (STAI-6). Secondary outcome measures are pain and stress levels, both measured with a Visual Analogue Scales (VAS), and well-being, measured with the Well-Being Numerical Rating Scales (WB-NRSs). The scales will be applied before and after each intervention.

This study seeks to contribute to improving mental health, wellbeing, and quality of care of patients and caregivers in the waiting area of the emergency units. This is the first study in Colombia investigating the effect live music therapy and pre-recorded music interventions in the emergency department.

DETAILED DESCRIPTION:
Main objective:

To determine the effect of standard care+ EMT or pre-recorded music on the state-anxiety, stress, pain, and wellbeing levels of anxiety-state, stress, pain, and well-being in adult patients and in the emergency waiting rooms of the Clínica Keralty Ibagué and Clínica Iberoamérica as compared to standard care alone.

Secondary objectives:

* Compare the sociodemographic and clinical characteristics of study participants according to the assigned intervention group.
* Evaluate the effect of EMT and pre-recorded music compared to the control group on state anxiety, stress, and wellbeing levels in adult patients and caregivers/companions in the emergency waiting rooms.
* Evaluate the effect of EMT and pre-recorded music compared to the control group on pain levels in patients in the emergency waiting rooms.
* Determine the variables that modify the effect of the interventions on primary and secondary outcomes in adult patients and their caregivers/companions in the emergency waiting rooms.

Methods Study Design

This study is a ramdomized clinical trial, multi-center, and pragmatic with three parallel arms - open label:

* Intervention Group 1 (GI1): Standard care + EMT
* Intervention Group 2 (GI2): Standard care + pre-recorded music
* Control Group (CG): Standard care alone

Study participants Study participants are adult patients and caregivers/companions in the emergency waiting room of both hospitals.

Concealment The concealment of the random assignment will be guaranteed using sealed, sequentially numbered, and opaque envelopes. The carbon paper inside the envelope will transfer the details of the random number and the group to which it is assigned (A, B or C). The envelopes will be sealed with tamper-proof security tape and opened sequentially on each day of intervention. The envelopes will be kept in a folder that will be kept on a locked shelf inside each clinic, which will be in custody by the research assistant at each participating clinic. The envelope will be opened 10 minutes before the start of the intervention to give the music therapists time to organize their equipment and instruments.

ELIGIBILITY:
Inclusion Criteria:

* Patients and caregivers/companions of legal age present in the emergency waiting room present during the intervention and control conditions.
* Patients whose triage does not represent immediate threat to life or severely ill patients (i.e., triage 3, 4 and 5)
* Patients and caregivers/companions with literacy skills.

Exclusion Criteria:

* Patients and caregivers/companions who report having hearing problems
* Patients and caregivers/companions with difficulties in understanding and/or filling out the questionnaires.
* Patients and/or caregivers/companions who do not consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 243 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
State-anxiety | The intervention will have a duration of twenty minutes. The STAI-6 will be administered prior to the intervention and immediately following its conclusion.
  It will be measured with the Spanish version of the state scale of the six-item State-Trait Anxiety Inventory (STAI-6) scored on a Likert scale from 1 "absence of anxiety" to 4 "high anxiety".

SECONDARY OUTCOMES:
Stress | The intervention will have a duration of twenty minutes. The VAS-S will be administered prior to the intervention and immediately following its conclusion.
  Stress levels will be measured by the Visual Analogue Stress Scale (VAS-S). The VAS-S consists of a 10-centimeter line divided into 10 points, each separated by 1 centimeter. 0 means the complete absence of stress and 10 the maximum possible stress. A cut-off of 7 points has been established as a significant stress level.
Pain (patients only) | The intervention will have a duration of twenty minutes. The VAS-P will be administered prior to the intervention and immediately following its conclusion.
  Perceived pain levels by patients will be measured with the Visual Analogue Pain Scale (VAS-P) consisting of a line of 10 centimeters divided into 10 points, each separated by 1 centimeter, where 0 means complete absence of pain and 10 the maximum possible pain.
Wellbeing | The intervention will have a duration of twenty minutes. The WB-NRS will be administered prior to the intervention and immediately following its conclusion.
  Well-being will be measured by the Well-being Numerical Rating Scales (WB-NRSs) consisting of a line divided into numbers from 1 to 10, where 1 indicates a state of absolute distress, and 10 a state of absolute well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ettenberger, PhD, Principal Investigator — keralty
Locations (2):
- Colombia (2):
  - Clínica Iberoamérica, Barranquilla, Atlántico
  - Clínica Keralty Ibagué, Ibagué, Tolima Department

IPD SHARING:
Plan to Share IPD: No
When the study ends, individual participant data could be shared with the approval of the research ethics committee.

REFERENCES:
- [Derived] Hernandez A, Diaz AM, Moreno OF, Suarez R, Amarillo M, Moreno AM, Rios Suarez BA, Gomez Gonzalez LM, Cristancho Olaya GA, Ettenberger M. Effect of Live Environmental Music Therapy and Prerecorded Music on State Anxiety, Stress, Pain, and Well-Being Levels of Patients and Caregivers in the Emergency Department Waiting Room: Protocol for a Multicenter Randomized Clinical Trial. JMIR Res Protoc. 2025 Jun 18;14:e69131. doi: 10.2196/69131. PMID 40531567